CLINICAL TRIAL: NCT03884712
Title: The Use of the CalmiGo Handheld Device in the Management of Patients With Anxiety and Panic Attack Symptoms in the Emergency Department
Brief Title: Using CalmiGo to Manage Anxiety and Panic Attack Symptoms in the Emergency Department
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yves Duroseau (Other)
Collaborators: Dendro Technologies, Inc (Unknown)
Responsible Party: Sponsor-Investigator, Yves Duroseau, Chairman of Emergency Medicine, Lenox Hill Hospital, Northwell Health
Organization: Northwell Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0033
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-09

CONDITIONS: Anxiety; Panic Attacks
Keywords: anxiety symptoms; panic attack symptoms; emergency department; CalmiGo
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CalmiGo Recipients (Experimental): This arm will receive a CalmiGo handheld device during their participation in the study. Participants will first complete validated surveys assessing their anxiety and panic attack symptoms. Investigators will then demonstrate how to use the CalmiGo handheld device. Participants will use the device with the investigator and then participants will use the device on their own for at least 2 times. After using CalmiGo, participants will complete validated surveys reassessing their anxiety and panic attack symptoms, asking about their past medical history, and inquiring about their experience using CalmiGo.
  Interventions: Device: CalmiGo

INTERVENTIONS:
Device: CalmiGo — The CalmiGo handheld device is a device of similar size to an inhaler that uses guided breathing, aromatherapy and grounding techniques to regulate breathing to bring users a sense of calm and relaxation. The CalmiGo handheld device is being tested in this study to alleviate participants' anxiety and panic attack symptoms.
  Other Names: myReLeaf

SUMMARY:
Currently, there are limited options in the management of anxiety and panic attack symptoms in the Emergency Department (ED). The most common treatment method is the use of anti-anxiety and anti-depressant medications; however, these drugs have serious health risks which make them ineffective as a long-term treatment option. The CalmiGo handheld device, formerly known as "myReLeaf", provides an alternative early intervention option in treating patients presenting with anxiety and panic attack symptoms by using guided breathing, aromatherapy, and grounding techniques. The hypothesis of this study is that CalmiGo will provide a drug-free, early intervention, and long-term treatment option in the ED that will improve patients' anxiety and panic attack symptoms.

Patients who present to the ED with anxiety or panic attack symptoms will be considered eligible for this study. These patients will be approached, and they will give informed consent to participate in the study. Patients will be enrolled in the study which consists of completing validated surveys asking about their anxiety and panic symptoms, using CalmiGo, and allowing investigators to access their medical records. These surveys will be completed before and after using CalmiGo in the ED to measure the presence and severity of anxiety and panic symptoms. The goal of this study is to analyze the effectiveness of using CalmiGo to improve anxiety and panic attack symptoms based on validated survey responses.

Overall, this study seeks to identify CalmiGo as an effective and alternative early intervention treatment option for patients presenting to the ED with anxiety or panic attack symptoms.

DETAILED DESCRIPTION:
Generalized Anxiety-the display of excessive anxiety or worry for months-is associated with several anxiety-related symptoms including restlessness, feeling wound-up or on edge, being easily fatigued, difficulty concentrating, having the mind go blank, irritability, muscle tension, difficulty controlling worry, and sleep abnormalities [The National Institute]. Panic attacks-sudden periods of intense fear-include symptoms of palpitations, pounding heart, accelerated heart rate, sweating, trembling, shaking, sensations of shortness of breath, smothering, choking, and feelings of impending doom. Panic attacks are symptoms of Panic Disorder-an anxiety disorder with reoccurring and unforeseen episodes of panic attacks [The National Institute].

Typically, treatment consists of a combination of psychotherapy, Cognitive Behavioral Therapy (CBT), support groups, stress-management techniques, and anti-anxiety and/or anti-depressant medications. The caveat with these treatment options is that only anti-anxiety or anti-depressant medications are available as an early intervention option, especially in the ED. The use of anti-anxiety and anti-depressant medications in the treatment of Generalized Anxiety, panic attacks, and Panic Disorder in the ED provides challenges on multiple levels. For instance, some anti-depressants now carry a "black box warning" from the U.S. Food and Drug Administration making these drugs high risk with potentially serious health consequences. Therefore, the limited treatments options for the symptoms of Generalized Anxiety, panic attacks, and Panic Disorder in the ED raises the need for alternative, early intervention treatments.

This research study aims to use the CalmiGo handheld device in the ED to aide in the short term and long term care of patients presenting with anxiety and panic attack symptoms. The standard of care for treating anxiety and panic attack symptoms in the ED consists of CBT, anti-anxiety medications such as benzodiazepines, and referring patients for a psychiatry consult, if appropriate. Compared to current treatment options in the ED, CalmiGo is a relatively less expensive, longer acting, drug-free device that addresses many distress related symptoms of anxiety through a combination of exhalation prolongation, aromatherapy, and grounding techniques [CalmiGo]. This study does not aim to eliminate the need for medication or other combination therapies; however, CalmiGo can provide an alternative treatment option that can alleviate clinical presentations of anxiety and panic symptoms and can be used as an early intervention treatment option.

This study will be conducted through the administration of validated surveys, teaching the participating subject how to use the CalmiGo device, and letting patients use the CalmiGo device on their own.

Two screening tools that have been clinically shown to be effective forms of assessing Generalized Anxiety, panic attacks, and Panic Disorder will be used to assess patients' anxiety and panic attack symptoms: the Generalized Anxiety Disorder subscale (GAD-7) and the Panic Symptom Scale (PSS). The GAD-7 uses a 7-item anxiety scale as a quick and easy tool to identify patients with anxiety and to monitor treatment response [Spitzer], [Ebell]. Whereas the GAD-7 is self-reporting, the PSS is an interview-based scale to determine the severity of 13 different panic symptoms as outlined by the DSM-IV [Locke], [Fleet]. The two of these screening tools are able to provide a thorough evaluation of patient's anxiety and panic attack symptoms.

Two other surveys will be conducted in order to gain demographic information including past medical history (Patient Demographic Survey) and a survey asking about the patient's experience with the CalmiGo device (CalmiGo questionnaire). These surveys have been designed by the study team.

To identify potentially eligible patients, investigators will screen the arrival board in the ED for specific chief complaints including anxiety, panic, non-cardiac chest pain (NCCP), unexplained chest pain (UCP), shortness of breath (SOB), and/or palpitations. Investigators will open the patient's electronic medical record to determine if patients are presenting to the ED with anxiety or panic attack symptoms, and investigators will ensure that the patient doesn't meet any exclusion criteria. Investigators will confirm with the patient's provider that the patient is experiencing anxiety and panic attack symptoms before approaching the patient about this study.

Investigators will approach the patient and obtain informed consent before enrolling the patient into the study.

First, the investigator will have the patient complete the GAD-7 and PSS surveys.

Following these surveys, the investigator will begin the CalmiGo device demonstration. The investigator will explain how the device works, what comes in the CalmiGo package, and will show the patient how to use CalmiGo by turning the device on and explaining the different commands of the device.

Then, the patient will use CalmiGo once for 3 minutes with the investigator is in the room to make sure that the patient understands how to use the device. The investigator will leave the patient for 20 minutes to let them use the CalmiGo device on their own. In these 20 minutes, the patient will be instructed to use CalmiGo for at least 2 additional times for 3 minutes each time. Once the investigator returns, the investigator will interview the patient with the PSS interviewed survey, the Patient Demographic Survey, and the CalmiGo questionnaire.

The investigator will input the data from the surveys completed during enrollment into REDCap, a HIPAA compliant database. The completed paper version of the surveys will be stored in a binder in a labeled locked cabinet at Lenox Hill Hospital.

Subjects will leave with a CalmiGo device along with user guides, a copy of their consent form and an additional aromatherapy element from the CalmiGo device.

Lastly, investigators will complete the Data Abstraction sheet after patients have been enrolled in the ED, completed all surveys and used the CalmiGo handheld device. Patients' medical charts will be accessed and reviewed to document the metrics on the Data Abstraction sheet, which will be completed on REDCap; there will be no paper documentation of the sheet. Abstracted information will include the patients' treatment in the ED, ED diagnosis, and ED disposition.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the LHH Emergency Department (ED)
* Presenting with anxiety and panic attack symptoms (confirmed by ED provider)
* Able to provide informed consent
* Must be aged 18 years or older

Exclusion Criteria:

* Pregnant patients
* Patients less than 18 years of age
* Prisoners
* Cognitively impaired.
* Asthma
* Chief obstructive pulmonary disorder (COPD)
* Bi-polar disorder
* Psychosis or delusional disorders
* History of substance abuse or dependence
* History of being suicidal
* Organic mental disorder
* Severe unstable medical illness
* Chronic respiratory disease
* History of seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in presentation and severity of anxiety and panic symptoms | 1 year
  Panic Symptom Scale (PSS) survey responses before using CalmiGo will be compared to the PSS survey responses after using CalmiGo. The PSS rates the severity of 13 panic symptoms on a scale of 0 to 4; a rating of 0 indicates that the symptom is not present and a rating of 4 indicates that the symptom is extremely severe. The sum of all the ratings for the 13 symptoms on the PSS (raw score) represents the overall severity of the patient's panic state. A lower raw score indicates a lesser severity of symptoms and a higher raw score indicates a higher severity of symptoms. If a patients raw score decreases after using CalmiGo, this would indicate an improvement in anxiety and panic attack symptoms and would indicate the effectiveness of using CalmiGo to treat anxiety and panic attack symptoms.

SECONDARY OUTCOMES:
Change in presentation and severity of anxiety and panic attack symptoms between patients who use and patients who do not use medications to treat anxiety or panic attacks | 1 year
  In the Patient Demographic Survey, participants will be asked if they use any medications to treat their anxiety or panic attack symptoms. In addition, the participants' electronic medical records will be reviewed for any anti-anxiety or panic attack medications. This will establish two cohorts of participants: those who use anti-anxiety and panic attack medications and those who do not. Changes in PSS survey responses from before using CalmiGo to after using CalmiGo will be compared between these cohorts to assess the effectiveness of CalmiGo to treat anxiety and panic attack symptoms in conjunction with anti-anxiety and panic attack medications. If the overall raw score for patients who uses anti-anxiety and panic attack medications decreases after using CalmiGo more than for patients who do not use medications, this would indicate that CalmiGo and medications benefit patients in reducing their anxiety and panic attack symptoms more than using CalmiGo on its own.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Duroseau, MD, Principal Investigator — Lenox Hill Hospital
Locations (1):
- Lenox Hill Hospital, Manhattan, New York, United States

REFERENCES:
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Ebell MH. Diagnosis of anxiety disorders in primary care. Am Fam Physician. 2008 Aug 15;78(4):501-2. No abstract available. PMID 18756659
- [Background] Fleet R, Foldes-Busque G, Gregoire J, Harel F, Laurin C, Burelle D, Lavoie K. A study of myocardial perfusion in patients with panic disorder and low risk coronary artery disease after 35% CO2 challenge. J Psychosom Res. 2014 Jan;76(1):41-5. doi: 10.1016/j.jpsychores.2013.08.003. Epub 2013 Aug 15. PMID 24360140
- [Background] Locke AB, Kirst N, Shultz CG. Diagnosis and management of generalized anxiety disorder and panic disorder in adults. Am Fam Physician. 2015 May 1;91(9):617-24. PMID 25955736
- See also: The National Institute of Mental Health. "Anxiety Disorders". The National Institute of Mental Health, U.S. Department of Health and Human Services. — https://www.nimh.nih.gov/health/topics/anxiety-disorders/index.shtml
- See also: CalmiGo. "The Science Behind CalmiGo". — https://calmigo.com/pages/the-science-behind-calmigo